CLINICAL TRIAL: NCT01669057
Title: Case-control Study on Environmental and Genetic Factors of Congenital Heart Disease
Brief Title: Study on Clinical Prognosis, Risk Factors and Genetic Basis of Congenital Heart Disease
Acronym: SCPRFGBCHD
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Ningbo Women & Children's Hospital (Other); Changzhou Maternal and Child Care Hospital (Other); Maternal and Child Health Hospital of Taian (Unknown); Maternal and Child Health Hospital of Wuxi (Unknown); Kunshan City Maternal and Child Health (Other); The First Affiliated Hospital of Xiamen University (Other); Maternal and Child Health Hospital, Jiading District (Other); Minhang Maternal and Children Health Care Hospital (Other)
Responsible Party: Principal Investigator, Guoying huang, Professor,President, Children's Hospital of Fudan University
Other Study IDs: KY2011-366
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; DNA variation; methylation; risk factors; supplements
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Congenital heart defect（CHD） group
- Normal control group

SUMMARY:
The objective of this study is to investigate the effect of parental peri-natal environmental risk factors and genetic factors on the development of Congenital Heart Disease (CHD). Our hypothesis is that the distributions of some environmental and genetic risk factors significantly differ between neonates with and without CHD.

DETAILED DESCRIPTION:
Congenital heart defect (CHD) is one of birth defects in the structure of the heart and/or great vessels. Many types of heart defects exist, most of which either obstruct blood flow in the heart or vessels near it, or cause blood to flow through the heart in an abnormal pattern. Heart defects are the leading cause of birth defect-related infant deaths. So far people recognize that the causes of CHD are the conjunct effect of environment and genetic factors, both of which remain unclear. The current stud aims at investigating all the possible perinatal parental environmental risk factors and underlying genetic factors to CHD, including DNA variation and methylations. A hospital-based 1:1 matched case control study is conducted. Subjects were recruited through neonatal screening program, which includes a clinical symptom screening followed by a cardiac ultrasound diagnosis for those with at least one clinical indicator. The blood sample of participant will be collected and the parents of subjects will be interviewed to completed a questionnaire including general information and possible risk factors to CHD.

ELIGIBILITY:
case group

Inclusion Criteria:

* Han ethnic
* 0~3 years old
* screened by 7 indicator, diagnosed by ultrasound

Exclusion Criteria:

* with other brith defects
* with Patent Ductus Arteriosus (PDA) and Patent Foramen Ovale (PFO)

Control group

Inclusion Criteria:

* Han ethnic
* 0~3 years old
* without any of 7 screen indicator , without CHD heart palpitations and other complaints about heart disease, born in the same hospital with cases

Exclusion Criteria:

With other birth defects

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population is from two ongoing projects- "Key Clinical Research Project Sponsored by Ministry of Health Screening, evaluation and intervention of congenital heart disease in newborn infants(2010-239)" and "Health and Public Welfare Research Project Sponsored by Ministry of Health of China Screening and evaluation of congenital heart disease in children of under 3 years old in the countryside(20102006)"
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2011-10; Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
genome-wide DNA SNPs and methylations | delivery
  DNA sample from neonate blood
perinatal supplements and drug using | three months before pregnancy till delivery
  questionnaire including supplements and drug using for mother

SECONDARY OUTCOMES:
Life risk factors of mother | three months before pregnancy till delivery
  smoking, drinking, health, family history
Life risk factors of father | three months before pregnancy till delivery
  smoking, drinking, health, family history
gestational weeks | delivery
birth weight | delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China